CLINICAL TRIAL: NCT02117895
Title: A Prospective RCT Study of Distal Pancreatectomy Combined With Left Celiac Plexus Resection for Pancreatic Cancer at the Body and Tail
Brief Title: Left Celiac Plexus Resection for Pancreatic Cancer at the Body and Tail
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Professor and Chair,Department of Pancreatic & Hepatobiliary Surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCI002
Record Dates: First submitted 2014-04-10; First posted 2014-04-21 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Pancreatic Cancer
Keywords: Distal Pancreatectomy; Celiac Plexus; Resection; Pancreatic Cancer; Body and Tail
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreatectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pancreatectomy & celiac plexus resection (Experimental): Left celiac plexus resection will be performed besides standard distal pancreatectomy. Celiac plexus at the left side of aorta, between celiac trunk and superior mesenteric artery will be resected.
  Interventions: Procedure: Celiac plexus resection; Procedure: Pancreatectomy
- Pancreatectomy (Active Comparator): Standard distal pancreatectomy includes distal pancreatectomy, splenectomy, and regional lymph nodes resection for pancreatic cancer at the body and tail. Regional lymph nodes includes group 8, 10, 11, 18, 7, 9, 14, 15, according to the 2003 edition of lymph nodes group system defined by Japan Pancreas Society (JPS).
  Interventions: Procedure: Pancreatectomy

INTERVENTIONS:
Procedure: Celiac plexus resection — Celiac plexus at the left side of aorta, between celiac trunk and superior mesenteric artery will be resected.
  Arms: Pancreatectomy & celiac plexus resection
Procedure: Pancreatectomy — Standard distal pancreatectomy includes distal pancreatectomy, splenectomy, and regional lymph nodes resection for pancreatic cancer at the body and tail. Regional lymph nodes includes group 8, 10, 11, 18, 7, 9, 14, 15, according to the 2003 edition of lymph nodes group system defined by Japan Pancreas Society (JPS).

SUMMARY:
This is a prospective study of left celiac plexus resection for pancreatic cancer at the body and tail during standard distal pancreatectomy.

DETAILED DESCRIPTION:
Pancreatic cancer has a property of nerve invasion. Pancreatic cancer cells first invade the nerves within the pancreas, then reach to the retroperitoneal celiax plexus and ganglion. Previous studies have showed nerve invasion was a negative prognostic factor for pancreatic cancer. Celiac plexus was thought as one the sources of tumor recurrence, which also led to severe abdominal and back pain in pancreatic cancer patients. This study is performed to confirm whether left celiac plexus resection could improve survival and relieve pain of pancreatic cancer patients.

Subjects undergoing surgery will be randomized to standard distal pancreatectomy plus left celiac plexus resection versus standard distal pancreatectom. Subjects will be followed every two months for survivorship or death to assess pain, quality of life measures, and narcotic pain control usage. The primary endpoint of overall survival and the secondary endpoint of disease-specific free survival will be determined at two year post surgery.The other pre-specified outcome of pain control will be determined at one year post surgery.

Block randomization will be done using a computer generated sheet. All surgeries will be performed under general anesthesia with epidural analgesia. The surgery will be either performed by or under the direct supervision of pancreatic surgeons with experience in pancreas surgery. Operative time, blood loss, blood product replacement and all intraoperative details will be recorded in the proforma. Patients will be shifted postoperatively to the anesthesia care unit (PACU) for observation and subsequently to the recovery or high dependency ward once stabilized. Postoperative details including period of postoperative pancreatic fistula,postoperative haemorrhage,postoperative pancreatitis , hospital stay and other complications will be recorded. Postoperative mortality will be defined as 30-day mortality plus death before discharge after surgery.All collected data will be entered into a statistical software package for subsequent analysis

ELIGIBILITY:
Inclusion Criteria:

* Signed informed content obtained prior to treatment
* Age ≥ 18 years and ≤ 80 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* The pathological staging does not exceed the stage IIB
* The expected survival after surgery ≥ 3 months
* Tumor locates at the body and tail of the pancreas without distant metastasis
* No celiac trunk and superior mesenteric artery invasion by Loyer grading
* No operation contraindication

Exclusion Criteria:

* The pathological staging exceed the stage IIB
* Pancreatic cancer at the head of the pancreas
* Benign tumor at the body and tail of the pancreas
* Distant metastasis
* Severe important organ function impairment
* Active second primary malignancy or history of second primary malignancy within the last 3 years
* Pregnant or nursing women
* Human immunodeficiency virus (HIV)-positive patients
* Patients who are unwilling or unable to comply with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years

SECONDARY OUTCOMES:
Disease-specific, recurrence-free survival | 2 years

OTHER OUTCOMES:
Pain Control | 12 months
  Paint control will be assess by the Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Jun Yu, M.D., Principal Investigator — Principal Investigator
Locations (1):
- Xian-Jun Yu, Shanghai, China

REFERENCES:
- [Result] Egawa S, Toma H, Ohigashi H, Okusaka T, Nakao A, Hatori T, Maguchi H, Yanagisawa A, Tanaka M. Japan Pancreatic Cancer Registry; 30th year anniversary: Japan Pancreas Society. Pancreas. 2012 Oct;41(7):985-92. doi: 10.1097/MPA.0b013e318258055c. PMID 22750974
- [Result] Fujii Y, Ueda M, Yoshida K, Matsuo K, Takeda K, Morioka D, Tanaka K, Endo I, Togo S, Shimada H. [Standard surgery as part of the multidisciplinary treatment for pancreatic cancer]. Nihon Geka Gakkai Zasshi. 2006 Jul;107(4):177-81. Japanese. PMID 16878410
- [Result] Yamamoto M, Ohashi O, Saitoh Y. Japan Pancreatic Cancer Registry: current status. Pancreas. 1998 Apr;16(3):238-42. doi: 10.1097/00006676-199804000-00006. PMID 9548661
- [Result] Wyse JM, Carone M, Paquin SC, Usatii M, Sahai AV. Randomized, double-blind, controlled trial of early endoscopic ultrasound-guided celiac plexus neurolysis to prevent pain progression in patients with newly diagnosed, painful, inoperable pancreatic cancer. J Clin Oncol. 2011 Sep 10;29(26):3541-6. doi: 10.1200/JCO.2010.32.2750. Epub 2011 Aug 15. PMID 21844506